CLINICAL TRIAL: NCT05655676
Title: 89Zr-labeled NY008 PET Imaging in Patients
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Affiliated Hospital of Jiangnan University (Other)
Responsible Party: Principal Investigator, Chunjing Yu, Director, Affiliated Hospital of Jiangnan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: LS2020001
Record Dates: First submitted 2022-12-05; First posted 2022-12-19 (Actual); Last update posted 2022-12-19 (Actual); Status verified 2022-12

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 89Zr-NY008 (Experimental)
  Interventions: Drug: 89Zr-NY008

INTERVENTIONS:
Drug: 89Zr-NY008 — Patients will receive a tracer (5-10mg, IV) dose of 89Zr (2-3mCi) labelled NY008

SUMMARY:
This is a single arm study to evaluate the safety and biodistribution of 89Zr-labeled NY008 PET Imaging in patients with multiple myeloma

ELIGIBILITY:
Inclusion Criteria:

1. Older than 18 years old, male or female;
2. Patients diagnosed with relapsing or refractory multiple myeloma；
3. LVEF≥50%；
4. ECOG score 0~2；

Exclusion Criteria:

1. Life expectancy of less than 3 months;
2. Participated in other clinical research within 1 month;
3. Recovery from major trauma (including surgery) within 28 days prior to study treatment;
4. Patients with systemic or locally severe infections, or other serious coexisting diseases;
5. Patients with abnormal immune function or who have recently used immunosuppressive or potentiating agents including various vaccines;
6. Patients with autoimmune diseases, including rheumatoid arthritis;
7. Inadequate control of arrhythmias, including atrial fibrillation;
8. Uncontrolled hypertension;
9. Patients with allergies or allergies to any component of the imaging agent or antibody;
10. Patients who cannot undergo PET/CT imaging scan;
11. Syphilis, HBV, HCV, or HIV positive subjects;
12. Male and female subjects of reproductive age cannot take effective contraceptive measures;
13. Pregnant or lactating women;
14. Patients with a history of mental illness or related conditions;
15. Other subjects considered unsuitable by researchers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-05-25 (Actual); Primary Completion 2023-05 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
Evaluation of tissue distribution of 89Zr-NY008 | 7 days
  Biodistribution of 89Zr-NY008 evaluated by radioactive uptake values (standardized uptake values, SUVs) in various organs will be reported.

CONTACTS AND LOCATIONS:
Locations (1):
- Affiliated Hospital of Jiangnan University, Wuxi, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No